CLINICAL TRIAL: NCT03144713
Title: Randomized Trial Comparing the Efficacy and Safety of Terlipressin With Albumin Versus Midodrine With Albumin Versus Albumin Alone in Prevention of Paracentesis Induced Circulatory Dysfunction in Cirrhosis
Brief Title: Efficacy and Safety of Terlipressin With Albumin Versus Midodrine With Albumin Versus Albumin Alone in Prevention of Paracentesis Induced Circulatory Dysfunction in Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-10
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2017-05

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Terlipressin; Midodrine; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Terlipressin (Experimental): Terlipressin 1mg intravenous bolus at the onset of paracentesis and the remaining as 1 mg doses intravenous at 8 and 16 h after the first dose. ( total -3mg)
  Interventions: Drug: Terlipressin
- Midodrine (Active Comparator): Midodrine 7.5 mg thrice daily for 3 days.
  Interventions: Drug: Midodrine
- Standard Medical Therapy (Active Comparator): Albumin-8g/L of tap- one half of dose at beginning of tap and rest half after 6 hours of tapping.
  Interventions: Drug: Albumin

INTERVENTIONS:
Drug: Terlipressin — Terlipressin 1mg intravenous bolus at the onset of paracentesis and the remaining as 1 mg doses intravenous at 8 and 16 h after the first dose. ( total -3mg)
  Arms: Terlipressin
Drug: Midodrine — Terlipressin 1mg intravenous bolus at the onset of paracentesis and the remaining as 1 mg doses intravenous at 8 and 16 h after the first dose. ( total -3mg)
  Arms: Midodrine
Drug: Albumin — Albumin-8g/L of tap- one half of dose at beginning of tap and rest half after 6 hours of tapping.
  Arms: Standard Medical Therapy

SUMMARY:
* Study Population: Patients admitted or seen in Out Patient Department, Department of Hepatology, Institute of Liver and Biliary Sciences.
* Study Design: Prospective Open Labeled Randomized Controlled Trial.
* Study Period: January 2017 to December 2017
* Intervention- Subjects will be randomized to 3 groups
* All patients will receive Standard medical therapy - Albumin-8g/L of tap- one half of dose at beginning of tap and rest half after 6 hours of tapping.

Group A - Subjects will receive Terlipressin 1mg intravenous bolus at the onset of paracentesis and the remaining as 1 mg doses intravenous at 8 and 16 h after the first dose. ( total -3mg) Group B - Midodrine 7.5 mg TDS x 3 days Group C - Standard medical therapy only

* Monitoring and Assessment: Clinical evaluation will be done at regular intervals.
* Adverse Effects: Rise in blood pressure, arrthymias, hyponatremia and rarely cardiovascular side effects have been noted.
* Stopping Rule: Development of PICD, hypertension ( BP>160/90mmhg-JNC class II)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cirrhosis who undergo Large volume paracentesis (> 5L)
2. Patients with age from 18-75 years

Exclusion Criteria:

1. Renal failure ( Creatinine>1.5mg/dl)
2. Recent Gastrointestinal bleeding within 7 days
3. Spontaneous bacterial Peritonitis
4. Patients with Cardiovascular disease (Electrocardiogram, 2D Echo)
5. Systemic arterial hypertension ( >160/90mmhg) Presence of hepatocellular carcinoma or portal vein thrombosis, Budd chiari syndrome
6. Patients with active untreated sepsis
7. Pregnancy
8. Patients with hepatic encephalopathy
9. No use of drugs affecting systemic hemodynamic 3 days prior to enrollment
10. Refusal to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-05-28 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Paracentesis Induced Circulatory Dysfunction (PICD). | Day 6

SECONDARY OUTCOMES:
Number of hospital admission withing 28 days in all the 3 groups | 28 days
Development of Hyponatremia in all the 3 groups | Day 28
  Hyponatremia is defined as S.Na < 130 meq/dL.
Development of Hepatic Encephalopathy in all the 3 groups | Day 28
  Hepatic Encephalopathy defined as West Haven Grade > 1
Recurrence of ascites in all the 3 groups | Day 28
Development of Acute Kidney Injury in all the 3 groups | Day 28
  Acute Kidney Injury is defined as increase S.Creatinine by more than 0.3 mg/dL
Survival in all the 3 groups | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No